CLINICAL TRIAL: NCT02990091
Title: Traumatic Brain Injury Recovery With n-3 Highly Unsaturated Fatty Acids (HUFAs): A Biomarker-driven Approach
Brief Title: Derivatives of Omega-3 HUFA as Biomarkers of Traumatic Brain Injury
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit participants
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Ramon Diaz-Arrastia, Presidential Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 826109
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: TBI
Keywords: TBI; DHA; omega-3 highly unsaturated fatty acids; synaptamide
MeSH Terms: interventions — Fatty Acids, Omega-3; Omacor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1,000mg/day n-3 HUFA (Experimental): Subjects will take one capsule daily starting at study enrollment (within 24 hours of injury) for 14 consecutive days.
  Interventions: Drug: Omega 3 fatty acid
- 4,000 mg/day n-3 HUFA (Experimental): Subjects will take 2 capsules twice daily starting at enrollment (within 24 hours of injury) for 14 consecutive days.
  Interventions: Drug: Omega 3 fatty acid
- 1 capsule safflower seed oil (Placebo Comparator): Subjects will take 1 capsule daily starting at enrollment (within 24 hours of injury) for 14 consecutive days.
  Interventions: Dietary Supplement: Safflower seed oil
- 4 capsules safflower seed oil (Placebo Comparator): Subjects will take 2 capsules twice daily starting at enrollment (within 24 hours of injury) for 14 consecutive days.
  Interventions: Dietary Supplement: Safflower seed oil

INTERVENTIONS:
Drug: Omega 3 fatty acid — LOVAZA is an FDA approved drug that is lawfully marketed in the United States by GlaxoSmithKline. There is no intent to use the results of this study to support a change in the labeling or the advertising of the drug. The highest dose administered for the study is the recommended prescribed dose of LOVAZA, therefore not creating greater risk. The patient population and route of administration will not significantly increase the risk associated with the use of the product. We will be using this drug under an IND exemption.
  Other Names: LOVAZA
  Arms: 1,000mg/day n-3 HUFA; 4,000 mg/day n-3 HUFA
Dietary Supplement: Safflower seed oil — Safflower seed oil is a commonly used dietary supplement. It has been chosen to be used as a comparative to the LOVAZA because of its non-omega-3 fats. There will be no increased risk due to dosage, route of administration, or patient population.
  Arms: 1 capsule safflower seed oil; 4 capsules safflower seed oil

SUMMARY:
This is a Phase 2 clinical trial designed to obtain data on relationships between potentially therapeutic doses of n-3 HUFA (highly unsaturated fatty acids) and their bioactive molecular derivatives, synaptamide, 17-hydroxy-DHA, and D-series resolvins, on clinical outcomes after TBI.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55
2. Documented/ verified TBI
3. Ability to swallow study agent within 48h of injury
4. If a sexually active female who is able to get pregnant, must be already taking birth control (prescription contraception)
5. Visual acuity/ hearing adequate for testing
6. Fluency in English or Spanish
7. Ability to provide informed consent for themselves
8. Co-enrolled in PARC-TBI protocol (IRB protocol #825783) or TRACK-TBI (IRB protocol #825503)
9. GCS 13-15

Exclusion Criteria:

1. Unstable respiratory or hemodynamic status
2. Evidence of penetrating brain injury
3. Requirement for craniotomy or craniectomy
4. Evidence of serious infectious complications
5. Acute ischemic heart disease or abnormal heart rhythm
6. History of abnormality in liver function
7. History or evidence of active malignancy
8. History of diabetes
9. History of pre-existing neurologic disorder, such as dementia, uncontrolled epilepsy, multiple sclerosis, strokes, brain tumors, prior severe TBI, or other disorder that confounds interpretation neuropsychological results
10. History of pre-existing disabling Axis I psychiatric disorder, such as major depression, schizophrenia, bipolar disorder or dementia
11. Allergy to omega-3 fatty acid ethyl esters or any ingredient of the study agent.
12. Known allergy to Safflower seed oil or ragweed plants
13. Consumption of fish or seafood 3 or more times per week on average or regular administration of omega-3 supplements (e.g., cod liver oil, borage oil, fish oil or evening primrose oil) defined as an average of 250 mg/day of n-3 HUFAs, over the previous 3 months.
14. Pregnancy or breast-feeding
15. Prisoners or patients in custody
16. Allergy, hypersensitivity, or intolerance to fish oils or omega-3 fats which are found in fish.
17. Use of anticoagulant medications or aspirin more than once per week within the last three months
18. Enrollment in any concurrent research protocols that would interfere with participant safety or research data integrity.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2023-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Relationship of varying doses of n-3 HUFAs on blood levels of the following bioactive metabolites | 14 days consecutively
  Bioactive metabolites being looked at are: synaptamide (n-docosahexaenoylethanolamine), 17-hydroxy-DHA, and D-series resolvins and determine relationship of n-3 HUFAs on blood levels of indicators of neuroinflammatory damage including Brain Derived Neurotrophic Factor (BDNF) in humans over 14 days after TBI.

SECONDARY OUTCOMES:
Relationship of n-3 HUFA blood levels and clinical outcomes measured by the Glasgow Outcome Scale-Extended (GOSE) | 14 days consecutively
  Clinical outcomes will include functional outcomes and will be assessed by using the TBI Common Data Elements Outcome battery. The analysis will focus on the Glasgow Outcome Scale-Extended (GOS-E) an ordinal scale based on a structured questionnaire which is universally used in TBI clinical studies.
Evalute potential adverse events | 14 days consecutively
  Evaluate potential adverse side effects including gastrointestinal tolerance and adverse neurological outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Diaz-Arrastia, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No